CLINICAL TRIAL: NCT00566917
Title: A Randomised Controlled Trial of Transvaginal Mesh (PROLIFT) Versus Anterior Colporrhaphy in Anterior Vaginal Wall Prolapse
Brief Title: Comparison Between Transvaginal Mesh and Traditional Surgery for Pelvic Organ Prolapse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The regional agreement on medical training and clinical research (ALF) between Stockholm county council and Karolinska Institutet. (Unknown); The Swedish Society of Medicine (Other); Investigators meetings supported by Gynecare Scandinavia. (Unknown)
Responsible Party: Associate professor Daniel Altman, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TVM III-07
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2008-05

CONDITIONS: Vaginal Prolapse
Keywords: Vagina; Prolapse; Anterior vaginal wall prolapse
MeSH Terms: conditions — Uterine Prolapse; Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Anterior colporrhaphy (standardised)
  Interventions: Procedure: Anterior colporrhaphy
- 2 (Experimental): Anterior PROLIFT
  Interventions: Procedure: Anterior PROLIFT

INTERVENTIONS:
Procedure: Anterior colporrhaphy — Standardised colporrhaphy of the anterior vaginal wall
  Arms: 1
Procedure: Anterior PROLIFT — Transvaginal mesh surgery of the anterior vaginal wall
  Arms: 2

SUMMARY:
Pelvic organ prolapse is characterized by a lack of pelvic floor support causing the pelvic organs and vaginal walls to protrude. For decades, suture repair techniques have been the primary choice of surgical treatment when indicated.

Traditional surgical techniques are frequently associated with unsatisfying anatomical recurrence rates and it is plausible that inherently weak, or damaged, pelvic floor supportive tissues need to be reinforced by a permanent support to avoid the high rates of recurrences commonly described using traditional techniques. Over the years sporadic attempts have been made to introduce novel surgical techniques using a variety of biomaterials with varying success. Despite a lack of clinical safety data, or compelling clinical evidence demonstrating that it improves outcomes compared to traditional suture techniques, use of biomaterials in pelvic reconstructive surgery has become widespread in just a few years .

It is likely that biomaterials need to be "anchored" in tissues not afflicted by the disease, in order to provide the intended pelvic floor support. This has given rise to transvaginal surgical techniques using a transobturator approach passing the mesh through the arcus tendineous fascia pelvis, or the sacrospinous ligaments through a transgluteal approach. Short term data from concluded and on-going safety assessments of these techniques has provided promising results and satisfying clinical outcomes. The aim of the present study is to compare anterior mesh repair (PROLIFT®) with traditional suture repair in a randomised trial.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive years in the past (biologically or reproductive decision)
* Prolapse of the anterior vaginal wall ≥POPQ-stadium II
* Prolapse specific pelvic symptom
* Being able to make an informed consent on participation
* Physically and cognitive capable of participating in the required follow-up
* No other pelvic floor surgery performed at the time of anterior repair
* No exclusion criteria fulfilled

Exclusion Criteria:

* Previous or current pelvic organ cancer (regardless of treatment)
* Severe rheumatic disease
* Insulin treated diabetes mellitus
* Connective tissue disorders (SLE, Sjögrens syndrome, Marfans syndrome, Ehlers Danhlos, collagenosis, polymyositis eller rheumatic myalgia)
* Current systemic steroid treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Combined primary outcome measure: anatomical assessment according to the pelvic organ prolapse quantification system and prolapse specific symptom | One year

SECONDARY OUTCOMES:
Quality of life | One year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Altman, MD, Assoc. prof., Study Chair — Karolinska Institutet; Christian Falconer, MD, Assoc. prof., Study Director — Karolinska Institutet at Danderyd University Hospital; Daniel Altman, MD, Assoc. prof., Principal Investigator — Karolinska Institutet
Locations (53):
- Denmark (2):
  - Nyköbing Hospital, Nyköbing
  - Skejby Hospital, Skejby
- Finland (9):
  - Hyvinkää Hospital, Hyvinkää
  - Jorvi Hospital, Jorvi
  - Central Finland Central Finland, Jyväskylä
  - Central Finland Central Hospital, Kotka
  - South Carelian Central Hospital, Lappeenranta
  - Lohja Hospital, Lohja
  - Porvoo Hospital, Porvoo
  - Lapland Central Hospital, Rovaniemi
  - Åbo Hospital, Turku
- Norway (15):
  - Akershus University Hospital, Ahus
  - Haukeland Hospital, Bergen
  - Innlandet Hospital, Brumunddal
  - Bærum Hospital, Bærum
  - Sörlandet Hospital, Flekkefjord
  - Förde Hospital, Förde
  - Ringerike Hospital, Hönefoss
  - Kongsberg Hospital, Kongsberg
  - Levanger Hospital, Levanger
  - Namsos Hospital, Namsos
  - Rikshospitalet, Oslo
  - Telemark Hospital, Skien
  - Stavanger University Hospital, Stavanger
  - The Regional Hospital in Tromsø, Tromsø
  - St Olav Hospital, Trondheim
- Sweden (27):
  - Borås Hospital, Borås
  - Höglandssjukhuset, Eksjö
  - Sahlgrenska Hospital, Gothenburg
  - Halmstad Hospital, Halmstad
  - Huddiksvall Hospital, Huddiksvall
  - Karlskoga Hospital, Karlskoga
  - Karlskrona Hospital, Karlskrona
  - Karlstad Hospital, Karlstad
  - Kristiansstad Hospital, Kristiansstad
  - Linköping University Hospital, Linköping
  - Sunderby Hospital, Luleå
  - Vrinnevi Hospital, Norrköping
  - Capio Läkargruppen Örebro, Örebro
  - Örebro University Hospital, Örebro
  - Skaraborg Hospital Skövde, Skövde
  - Södertälje Hospital, Södertälje
  - Danderyd University Hospital, Stockholm
  - Karolinska University Hospital Huddinge, Stockholm
  - S:t Göran Hospital, Stockholm
  - South Hospital, Stockholm
  - Sundsvall Hospital, Sundsvall
  - NÄL Hospital, Trollhättan
  - Uppsala Academic Hospital, Uppsala
  - Värnamo Hospital, Värnamo
  - Västerås Hospital, Västerås
  - Västervik Hospital, Västervik
  - Ystad Hospital, Ystad

REFERENCES:
- [Derived] Baessler K, Christmann-Schmid C, Haya N, Mowat A, Chen Z, Wallace SA, Yeung E, Maher C. Surgery for women with pelvic organ prolapse with or without stress urinary incontinence. Cochrane Database Syst Rev. 2026 Feb 6;2(2):CD013108. doi: 10.1002/14651858.CD013108.pub2. PMID 41649019
- [Derived] Yeung E, Baessler K, Christmann-Schmid C, Haya N, Chen Z, Wallace SA, Mowat A, Maher C. Transvaginal mesh or grafts or native tissue repair for vaginal prolapse. Cochrane Database Syst Rev. 2024 Mar 13;3(3):CD012079. doi: 10.1002/14651858.CD012079.pub2. PMID 38477494
- [Derived] Elmer C, Falconer C, Hallin A, Larsson G, Ek M, Altman D; Nordic Transvaginal Mesh Group. Risk factors for mesh complications after trocar guided transvaginal mesh kit repair of anterior vaginal wall prolapse. Neurourol Urodyn. 2012 Sep;31(7):1165-9. doi: 10.1002/nau.22231. Epub 2012 Apr 19. PMID 22517125
- [Derived] Altman D, Vayrynen T, Engh ME, Axelsen S, Falconer C; Nordic Transvaginal Mesh Group. Anterior colporrhaphy versus transvaginal mesh for pelvic-organ prolapse. N Engl J Med. 2011 May 12;364(19):1826-36. doi: 10.1056/NEJMoa1009521. PMID 21561348